CLINICAL TRIAL: NCT03913624
Title: 35 Hz Versus 50 Hz Frequency Stimulation Effects on Motor Recovery in Older Adults After Stroke. A Randomized Clinical Trial
Brief Title: Effectiveness of Neuromuscular Electrical Stimulation After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Trinidad Sentandreu-Mañó, Principal Investigator, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43/09
Record Dates: First submitted 2019-03-09; First posted 2019-04-12 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Stroke
Keywords: Rehabilitation; Electric stimulation; Upper limb; Aging
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

ARMS (3):
- 50 Hz NMES group (Experimental): Neuromuscular electrical stimulation (NMES) was applied on wrist and finger extensors for 30 minutes, 3 sessions per week for 8 weeks. The main electrostimulation parameters consisted of low-frequency current, a stimulation frequency of 50 Hz, symmetrical rectangular biphasic wave, and pulse duration of 300 μs.
  Interventions: Other: Neuromuscular electrical stimulation
- 35 Hz NMES group (Experimental): Neuromuscular electrical stimulation (NMES) was applied on wrist and finger extensors for 30 minutes, 3 sessions per week for 8 weeks. The main electrostimulation parameters consisted of low-frequency current, a stimulation frequency of 35 Hz, symmetrical rectangular biphasic wave, and pulse duration of 300 μs.
  Interventions: Other: Neuromuscular electrical stimulation
- Control group (No Intervention): Conventional treatment

INTERVENTIONS:
Other: Neuromuscular electrical stimulation
  Arms: 35 Hz NMES group; 50 Hz NMES group

SUMMARY:
A Randomized Clinical Trial (RCT) was conducted to determine the effects of two neuromuscular electrical stimulation protocols with different stimulation frequencies on motor recovery in older adults with spastic hemiparesis after a stroke.

DETAILED DESCRIPTION:
Impairment of the upper limb is one of the most frequent consequences of stroke and directly impacts on the patient's functional status and quality of life. It is estimated that less than 50% of stroke survivors will recover arm function, which will exert a great economic, social and personal toll.

Neuromuscular electrical stimulation (NMES) is one of the techniques suggested for upper limb recovery in stroke patients. However, after considering the bibliographic background, more studies are required in order to test its effectiveness, to establish the most efficient NMES protocols and to assess the characteristics of the patients who can benefit the most from this treatment. With this regard, the parameters of the stimulation are currently subject to debate, and more data are needed to optimize the application of this treatment. The aim of this study was to evaluate and compare the effects of two neuromuscular electrical stimulation protocols with different stimulation frequencies on motor impairment, kinaesthetic sensation, functional motor ability, activities of daily living, and quality of life in older adults with spastic hemiparesis suffering a stroke.

To cope with the objective of the present study, RCT was conducted. Subjects who met inclusion criteria were recruited from a hospital rehabilitation unit. After the screening and signed consent, participants were randomly allocated to the control group or one of both experimental groups. NMES was applied on wrist and finger extensors for 30 minutes, 3 sessions per week for 8 weeks. The electrostimulation protocols were only differentiated in the parameter of the stimulation frequency, 35 Hz or 50 Hz, depending on the experimental group to which the patient belonged to. Outcome measures were collected at the beginning, after 4 and 8 weeks of treatment, and after a follow-up period (4 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years
* Post-stroke spastic hemiparesis
* Mild-moderate hand impairment
* A score ≤ 3 on the modified Ashworth scale for wrist and finger flexors
* Active wrist extension ≥ 5º from the resting position
* Wrist extension response to stimulation
* Post-stroke period < 18 months
* Clinical stability
* Mini-Mental State Examination score ≥ 23

Exclusion Criteria:

* Previous hemiparesis due to stroke
* Dermatological reactions with the application of stimulation
* Significant sensory deficits in the affected arm
* Previous musculoskeletal problems of the hand
* Treatment with the botulin toxin
* Anti-spastic medication usage
* Cardiac pacemaker, implanted electronic device, or metal implants in the affected arm
* Complex regional pain syndrome
* Severe aphasia, history of epileptic seizures, psychiatric disorder or important alterations of behavior
* Severe visual impairment
* Any comorbid neurological disease
* Important deformity or obesity that affects the application of the NMES
* Potentially fatal cardiac arrhythmia or another decompensated heart disease
* Systemic infectious process, cancer or another terminal disease

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in range of motion | The groups were assessed at baseline and 12 weeks post-intervention.
  A universal goniometer was used to measure the resting angle, active extension and passive extension of the wrist. A special JAMAR finger goniometer was used to evaluate the resting angle and active extension of the metacarpophalangeal joints of the fingers.
Change in dynamometric strength | The groups were assessed at baseline and 12 weeks post-intervention.
  The grip strength was assessed by means of a JAMAR hydraulic hand dynamometer and the pinch strength using the JAMAR hydraulic pinch gauge. Unit of measurement was kgf. Three repetitions were done in both evaluations, taking the highest value and leaving a resting period of 1 minute between them.
Change in muscle tone | The groups were assessed at baseline and 12 weeks post-intervention.
  Hypertonia of the finger and wrist flexors was measured using the modified Ashworth scale (MAS). MAS was used to categorize the severity of muscle tone by judging resistance to passive movement. It is a 6-point scale (0, 1, 1+ 2, 3, and 4) that ranges from 1 (=no increase in tone) to 4 (=limb rigid in flexion or extension). The assessment was started 5 minutes after laying the subject down in the supine position and using a single passive movement to evaluate each muscle group.
Change in functional motor ability | The groups were assessed at baseline and 12 weeks post-intervention.
  Manual dexterity was assessed by Box and block test.

SECONDARY OUTCOMES:
Change in the mean electromyographic (EMG) amplitude | The groups were assessed at baseline and 12 weeks post-intervention.
  The Muscle Trainer model METR-0 (Mega Electronics Ltd, Kuopio, Finland) surface electromyograph was used. Circular adhesive surface bipolar electrodes (Ambú® Blue Sensor) were used and placed parallel to the muscle fibers. The mean amplitude of the EMG signal (in µV) of the muscle was recorded in the radial extensor and the radial flexor of the carpus. The patient was asked to perform maximum voluntary isometric contractions of both the flexors and extensors of the wrist for five seconds against manual resistance and the electrical activity of both the agonist and antagonist muscles was recorded simultaneously.
Change in the peak EMG amplitude | The groups were assessed at baseline and 12 weeks post-intervention.
  The Muscle Trainer model METR-0 (Mega Electronics Ltd, Kuopio, Finland) surface electromyograph was used. Circular adhesive surface bipolar electrodes (Ambú® Blue Sensor) were used and placed parallel to the muscle fibers. The peak amplitude of the EMG signal (in µV) of the muscle was recorded in the radial extensor and the radial flexor of the carpus. The patient was asked to perform maximum voluntary isometric contractions of both the flexors and extensors of the wrist for five seconds against manual resistance and the electrical activity of both the agonist and antagonist muscles was recorded simultaneously.
Change in the antagonist co-activation ratio | The groups were assessed at baseline and 12 weeks post-intervention.
  The Muscle Trainer model METR-0 (Mega Electronics Ltd, Kuopio, Finland) surface electromyograph was used. The antagonist co-activation ratio, both for the flexors and extensors of the wrist, was calculated using the following formula (antagonist activity/ [agonist activity + antagonist activity] x100%) (Reference: J Electromyogr Kinesiol. 2014;24:731-738) which provides an estimate of the relative activation of the agonist-antagonist muscle pair and also of the magnitude of the co-activation of the antagonist.
Change in kinaesthetic sensation | The groups were assessed at baseline and 12 weeks post-intervention.
  Hand kinaesthesia was assessed by the Revised Nottingham Sensory Assessment (RNSA) subscale. The RNSA includes three subscales: tactile sensation, kinesthetic sensation, and stereognosis. For kinesthetic sensation, all three aspects of the movement were tested: appreciation of movement, its direction, and accurate joint position sense. The limb on the affected side of the body was supported and moved by the examiner in various directions but the movement is only at one joint at a time. The patients were asked to mirror the change of movement with the other limb. This subscale ranges from 0 to 3. Higher scores indicate better kinaesthetic sensation.
Change in activities of daily living | The groups were assessed at baseline and 12 weeks post-intervention.
  A score of the Barthel Index ranging from 0 to 100 was collected where 0 is the minimum (worst outcome) and 100 is the maximum (best outcome).
Change in health-related quality of life | The groups were assessed at baseline and 12 weeks post-intervention.
  COOP/WONCA charts were used. This instrument is a generic health status questionnaire which comprises nine single-item scales: physical fitness, feelings (mental well-being), daily activities, social activities, change in health and overall health, pain, social support, and quality of life. Each chart is rated on a five-point Likert scale with accompanying pictorial representations. Lower scores indicate better health-related quality of life.

OTHER OUTCOMES:
Intervention costs | Intervention costs were recorded from the baseline to 12 weeks.
  Intervention costs related to staff, consumables, and capital for intervention were calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Trinidad Sentandreu Mañó, PT, PhD, Principal Investigator — University of Valencia; J. Ricardo Salom Terrádez, MD, PhD, Study Chair — Doctor Peset University Hospital; J. Manuel Tomas, PhD, Study Chair — University of Valencia
Locations (1):
- Doctor Peset University Hospital, Valencia, Spain